CLINICAL TRIAL: NCT05221918
Title: Comparison of CSF Flow Metrics Across MRI Platforms
Brief Title: A Study to Compare CSF Flow Metrics Across Platforms
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Petrice M. Cogswell, Principal Investigator, Mayo Clinic
Other Study IDs: 21-002907
Record Dates: First submitted 2022-01-23; First posted 2022-02-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research is to find out more about detecting movement of CSF (fluid around the brain) with MRI. Researchers are doing this research study to find out how measurements of CSF movement differ among MRI machines and how image quality is changed by reducing the scan time.

ELIGIBILITY:
Inclusion Criteria:

- A healthy volunteer will be defined as an otherwise healthy person who does not have a medical condition that affects brain function or have problems with concentration, memory, balance, or coordination.

Exclusion Criteria:

- Subjects with non-MRI compatible devices, required sedation (claustrophobia or unable to remain still for exam), or women who are pregnant will be excluded.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will include healthy young adults, ages 18-40 years.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Comparison of flow metrics among scanners | February -December 2022
  Flow metrics such as average total flow will be compared among multiple MRI scanners
Comparison of flow metrics between scans with and without parallel imaging | February -December 2022
  Flow metrics such as the average total flow will be compared between sequences acquired with and without acceleration techniques, including parallel imaging, for a given scanner

CONTACTS AND LOCATIONS:
Overall Officials: Petrice Cogswell, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States